CLINICAL TRIAL: NCT00543361
Title: A Double-Blind, Randomized, Active-Controlled MK0767 and Metformin Comparator Study in Type 2 Diabetic Patients Inadequately Controlled on Diet and Exercise
Brief Title: Study MK0767 and Metformin in Type 2 Diabetic Patients (0767-020)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0767-020; MK0767-020; 2007_627
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — MK0767

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0767 — Duration of Treatment: 52 Weeks
Drug: Comparator: placebo (unspecified) — Duration of Treatment: 52 Weeks
Drug: Comparator: metformin — Duration of Treatment: 52 Weeks

SUMMARY:
The purpose of the study is to assess how MK0767, compared to Metformin, performs in lowering blood glucose levels in patients whose Type II diabetes is not controlled by diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients are men and non-pregnant women ages 21 to 78 years
* Patients either not on antihyperglycemic medications (>8 weeks), or being treated with a single oral antihyperglycemic agent & willing to discontinue therapy for the duration of the study

Exclusion Criteria:

* Patient has history of type 1 diabetes mellitus and or history of ketoacidosis
* Patients undergoing surgery within 30 days of Visit 1
* Patients taking Warfin or Warfin-like anticoagulants
* Patients on a weight loss program with on-going weight loss or starting an intensive exercise program within 4 weeks of Visit 1/Week 9

Ages: 21 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2003-05; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
This study will assess the lipid lowering effectiveness of MK0767 compared to metformin over the course of 52 weeks. | over the course of 52 weeks

SECONDARY OUTCOMES:
MK0767 will be safe and well tolerated. | over the course of 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC